CLINICAL TRIAL: NCT05403203
Title: Prediction of Need of Blood Transfusion > 4 Units of Packed RBCS in Cases Diagnosed With Placenta Previa During Cesarean Section .
Brief Title: Prediction of Bleeding in Placenta Previa
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youssef khalaf makary, Principal investigator, Assiut University
Other Study IDs: bleeding in placenta previa
Record Dates: First submitted 2022-05-11; First posted 2022-06-03 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-05

CONDITIONS: Placenta Previa Bleeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the ability of clinical and sonographic variables to predict the need of blood transfusion > 4 units of packed RBCS in women undergoing cesarian section for placenta previa .

DETAILED DESCRIPTION:
Womenwith placenta previa after 32 weeks will be assessed for participation if they are eligible an adequate data will be taken :

- Clinical factors : including maternal age, abortion history, cesarean section history, gestational age at delivery, whether the operation will be carried out as an emergency surgery, and whether bleeding has started before the operation, will evaluated. The number of abortion history will be counted only if a dilatation and curettage was performed. Preoperative hemoglobin and hematocrit values will be checked. The amount of PRBCs transfused during operation will be measured.

-Ultrasonographic factor: Adiagnosis of placenta previa was made when the placenta covered the internal orifice of the cervix after 32 weeks' gestation. We will check for the presence of a hypoechoic area between the myometrium and the placenta. The vascularity of the placenta will be classified as normal or hypervascular on color Doppler imaging. We will examine the location of placenta ( anterior . posterior. Anterior with lateral deviation. Posterior with lateral deviation) and presence ofintraplacental lacunae (an irregular area of low echogenicity larger than 1 cm × 1 cm in the placental parenchyma)

* Intraoperative factor:

Assess surgeon years of experience Management plan hemostatic sutures other conservative management hysterectomy (primary or secondary) Assessment of amount of blood taken in 24 h from operation

ELIGIBILITY:
Inclusion Criteria:

* women with placenta previa after 32 weeks
* women with placenta accreta after 32 weeks

Exclusion Criteria:

* abruption placenta
* unavilable or limited avilability of blood group

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: women with placenta previa or accreta after 32 weeks
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Ability of a score of the study to predict the need for blood transfusion > 4 units of packed RBCs | baseline
  It is a questionnaire Data collection of full personal history and obstetric and gynocological history and sonographic data . The data will be collected and entered on Microsoft access data base to be analysed using the Statistical Package for Social Science (SPSS Inc. ,Chicago,version 21) groups difference will be assessed by independent sample t-test and Chi square for prediction of receiving >4 units 0f packed RBCS will be assessed by logistic Regression then a scoring system of factors that will prove independently significant . The predictive accuracy of the scoring system will be analysed using ROC curve

SECONDARY OUTCOMES:
The effect on morbidity of pregnant women . | baseline
  Morbidities were defined as organ system dysfunctions related to severe obstetric hemorrhage and included: acute respiratory distress syndrome (impairment of respiratory function needing ventilation, oxygen supplementation, or decreased physical activity level as compared to pre-pregnancy), cerebral impairment (seizures, unconsciousness, or cognitive/motor loss), renal failure (creatinine > 1.5 mg/dL or increased >1.0 mg/dL above baseline, oliguria; <120 mL output in 4-hour intervals), and heart failure (impairment of cardiac function according to New York Heart Disease Classification)
The effect on mortality of pregnant women . | Baseline

REFERENCES:
- [Background] Silver RM. Abnormal Placentation: Placenta Previa, Vasa Previa, and Placenta Accreta. Obstet Gynecol. 2015 Sep;126(3):654-668. doi: 10.1097/AOG.0000000000001005. PMID 26244528
- [Background] Rouse DJ, MacPherson C, Landon M, Varner MW, Leveno KJ, Moawad AH, Spong CY, Caritis SN, Meis PJ, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai BM, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Blood transfusion and cesarean delivery. Obstet Gynecol. 2006 Oct;108(4):891-7. doi: 10.1097/01.AOG.0000236547.35234.8c. PMID 17012451
- [Background] Silver RM, Branch DW. Placenta Accreta Spectrum. N Engl J Med. 2018 Apr 19;378(16):1529-1536. doi: 10.1056/NEJMcp1709324. No abstract available. PMID 29669225
- [Background] Dahlke JD, Mendez-Figueroa H, Maggio L, Hauspurg AK, Sperling JD, Chauhan SP, Rouse DJ. Prevention and management of postpartum hemorrhage: a comparison of 4 national guidelines. Am J Obstet Gynecol. 2015 Jul;213(1):76.e1-76.e10. doi: 10.1016/j.ajog.2015.02.023. Epub 2015 Feb 28. PMID 25731692
- [Background] Weiniger CF, Elram T, Ginosar Y, Mankuta D, Weissman C, Ezra Y. Anaesthetic management of placenta accreta: use of a pre-operative high and low suspicion classification. Anaesthesia. 2005 Nov;60(11):1079-84. doi: 10.1111/j.1365-2044.2005.04369.x. PMID 16229692
- [Background] Snyder CW, Weinberg JA, McGwin G Jr, Melton SM, George RL, Reiff DA, Cross JM, Hubbard-Brown J, Rue LW 3rd, Kerby JD. The relationship of blood product ratio to mortality: survival benefit or survival bias? J Trauma. 2009 Feb;66(2):358-62; discussion 362-4. doi: 10.1097/TA.0b013e318196c3ac. PMID 19204508
- [Background] Pacheco LD, Saade GR, Costantine MM, Clark SL, Hankins GD. An update on the use of massive transfusion protocols in obstetrics. Am J Obstet Gynecol. 2016 Mar;214(3):340-4. doi: 10.1016/j.ajog.2015.08.068. Epub 2015 Sep 5. PMID 26348379
- [Background] Finberg HJ, Williams JW. Placenta accreta: prospective sonographic diagnosis in patients with placenta previa and prior cesarean section. J Ultrasound Med. 1992 Jul;11(7):333-43. doi: 10.7863/jum.1992.11.7.333. PMID 1522623
- [Background] Farquhar CM, Li Z, Lensen S, McLintock C, Pollock W, Peek MJ, Ellwood D, Knight M, Homer CS, Vaughan G, Wang A, Sullivan E. Incidence, risk factors and perinatal outcomes for placenta accreta in Australia and New Zealand: a case-control study. BMJ Open. 2017 Oct 5;7(10):e017713. doi: 10.1136/bmjopen-2017-017713. PMID 28982832
- [Background] Gibbins KJ, Einerson BD, Varner MW, Silver RM. Placenta previa and maternal hemorrhagic morbidity. J Matern Fetal Neonatal Med. 2018 Feb;31(4):494-499. doi: 10.1080/14767058.2017.1289163. Epub 2017 Feb 21. PMID 28140723